CLINICAL TRIAL: NCT07030868
Title: A Phase 2, Parallel-Group, Double-Blind 4-arm Study to Investigate the Effects of Treatment With LY3549492 Tablets Compared With Placebo in an Obese or Overweight Population With Type-2 Diabetes (T2D)
Brief Title: A Study of LY3549492 in Adults With Obesity or Overweight With Type 2 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated for strategic business reasons
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27321; W8M-MC-GN02 (Other: Eli Lilly and Company); W8M-MC-CWMM (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Overweight; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3549492 Dose 1 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY6249492
- LY3549492 Dose 2 Fast Titration (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY6249492
- LY3549492 Dose 2 Slow Titration (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY6249492
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY6249492 — Administered orally
  Arms: LY3549492 Dose 1; LY3549492 Dose 2 Fast Titration; LY3549492 Dose 2 Slow Titration
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study, performed under the master protocol W8M-MC-CWMM (NCT06143956), is to evaluate the effects of treatment with LY3549492 compared to placebo in adult participants with obesity or who are overweight with type 2 diabetes.

Participation in the study will last about 11 months.

ELIGIBILITY:
Inclusion Criteria:

W8M-MC-GN02:

* Assigned male at birth
* Assigned female at birth, who are of non-childbearing potential
* Have type 2 diabetes

W8M-MC-CWMM:

* Have a BMI ≥27 kilograms per square meter (kg/m²)
* Have had a stable body weight for the 3 months prior to randomization (<5% body weight gain and/or loss

Exclusion Criteria:

W8M-MC-GN02:

* Individuals who are of childbearing potential
* Have a history of acute or chronic pancreatitis
* Have any of the following cardiovascular conditions within 6 months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure.

W8M-MC-CWMM:

* Have a prior or planned surgical treatment for obesity, except prior liposuction or abdominoplasty, if performed >1 year prior to screening
* Have type 1 diabetes mellitus, latent autoimmune diabetes in adults, or history of ketoacidosis or hyperosmolar coma
* Have poorly controlled hypertension
* Have signs and symptoms of any liver disease other than nonalcoholic fatty liver disease
* Have a history of symptomatic gallbladder disease within the past 2 years
* Have a lifetime history of suicide attempts

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 32

SECONDARY OUTCOMES:
Change from Baseline in Body Weight | Baseline, Week 32
Percentage of Participants Who Achieve ≥5% Body Weight Reduction | Baseline, Week 32
Percentage of Participants Who Achieve ≥10% Body Weight Reduction | Baseline, Week 32
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 32
Pharmacokinetics (PK): Average Concentration of LY3549492 | Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (42):
- United States (38):
  - HOPE Research Institute, Phoenix, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - NorCal Medical Research, Inc, Greenbrae, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Medical Research Partners, Ammon, Idaho
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Knownwell, Needham, Massachusetts
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Headlands Research - Detroit, Southfield, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Clinvest Headlands Llc, Springfield, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Lucas Research, Inc., New Bern, North Carolina
  - Quality Medical Research, Nashville, Tennessee
  - IMA Clinical Research Austin, Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Tekton Research - Fredericksburg Road, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Spectrum Medical, Inc., Danville, Virginia
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
- Argentina (4):
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY3549492 in Adults With Obesity or Overweight With Type 2 Diabetes — https://trials.lilly.com/en-US/trial/619929